CLINICAL TRIAL: NCT03255291
Title: Communicating Multiple Disease Risks: A Translation of Risk Prediction Science
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 201706063; R01CA190391 (NIH)
Record Dates: First submitted 2017-08-07; First posted 2017-08-21 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned by a computer algorithm to one of six intervention arms according to a 3 (risk display format: text, table, ladder) x 2 (imagery behavior: exercise, sleep) between-subjects factorial design. Although randomization was done at the same time and at the beginning of the study, participants received the risk display intervention first, then answered a survey containing two of the primary outcomes, then received the mental imagery intervention followed by another survey.
Who Masked: Investigator
Masking Description: The research staff will be blinded to participants' risk display format conditions, but they will be unblinded to mental imagery behavior condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Risk Display Format:Risk Ladder:Imagery Behavior:Exercise (Experimental): * With help from a research assistant, participants complete the Risk Assessment App. The App asks demographic & health questions. It then provides personalized risk estimates for participants' current activity level & how it would change with regular exercise.
  * Participants take Baseline Survey 1.
  * Participants listen to an audio recording that guides them through a mental imagery activity. They write down an exercise goal & are asked to practice the mental imagery twice a day for 3 weeks.
  * Participants take Baseline Survey 2.
  * Participants receive text messages reminding them to practice the mental imagery twice daily for 5 minutes each time (3 texts a week for 3 weeks).
  * Participants take surveys via text at the end of each week for 4 weeks.
  * 90 days post-baseline, participants complete a survey sent through the mail.
  * Participants may be contacted for another survey 1 year later.
  Interventions: Behavioral: Risk Assessment App; Other: Surveys; Behavioral: Audio Recording - Exercise; Other: Text message reminders; Other: Text Message Survey
- Risk Display Format:Risk Ladder:Imagery Behavior:Sleep (Experimental): * With help from a research assistant, participants complete the Risk Assessment App. The App asks demographic & health questions. It then provides personalized risk estimates for participants' current activity level & how it would change with regular exercise.
  * Participants take Baseline Survey 1.
  * Participants listen to an audio recording that guides them through a mental imagery activity. They write down a sleep goal & are asked to practice the mental imagery twice a day for 3 weeks.
  * Participants take Baseline Survey 2.
  * Participants receive text messages reminding them to practice the mental imagery twice daily for 5 minutes each time (3 texts a week for 3 weeks).
  * Participants take surveys via text at the end of each week for 4 weeks.
  * 90 days post-baseline, participants complete a survey sent through the mail.
  * Participants may be contacted for another survey 1 year later.
  Interventions: Behavioral: Risk Assessment App; Behavioral: Audio Recording - Sleep; Other: Surveys; Other: Text message reminders; Other: Text Message Survey
- Risk Display Format:Table:Imagery Behavior:Exercise (Experimental): * With help from a research assistant, participants complete the Risk Assessment App. The App asks demographic & health questions. It then provides personalized risk estimates for participants' current activity level & how it would change with regular exercise.
  * Participants take Baseline Survey 1.
  * Participants listen to an audio recording that guides them through a mental imagery activity. They write down an exercise goal & are asked to practice the mental imagery twice a day for 3 weeks.
  * Participants take Baseline Survey 2.
  * Participants receive text messages reminding them to practice the mental imagery twice daily for 5 minutes each time (3 texts a week for 3 weeks).
  * Participants take surveys via text at the end of each week for 4 weeks.
  * 90 days post-baseline, participants complete a survey sent through the mail.
  * Participants may be contacted for another survey 1 year later.
  Interventions: Behavioral: Risk Assessment App; Other: Surveys; Behavioral: Audio Recording - Exercise; Other: Text message reminders; Other: Text Message Survey
- Risk Display Format:Table: Imagery Behavior:Sleep (Experimental): * With help from a research assistant, participants complete the Risk Assessment App. The App asks demographic & health questions. It then provides personalized risk estimates for participants' current activity level & how it would change with regular exercise.
  * Participants take Baseline Survey 1.
  * Participants listen to an audio recording that guides them through a mental imagery activity. They write down a sleep goal & are asked to practice the mental imagery twice a day for 3 weeks.
  * Participants take Baseline Survey 2.
  * Participants receive text messages reminding them to practice the mental imagery twice daily for 5 minutes each time (3 texts a week for 3 weeks).
  * Participants take surveys via text at the end of each week for 4 weeks.
  * 90 days post-baseline, participants complete a survey sent through the mail.
  * Participants may be contacted for another survey 1 year later.
  Interventions: Behavioral: Risk Assessment App; Behavioral: Audio Recording - Sleep; Other: Surveys; Other: Text message reminders; Other: Text Message Survey
- Risk Display Format:Text:Imagery Behavior:Exercise (Experimental): * With help from a research assistant, participants complete the Risk Assessment App. The App asks demographic & health questions. It then provides personalized risk estimates for participants' current activity level & how it would change with regular exercise.
  * Participants take Baseline Survey 1.
  * Participants listen to an audio recording that guides them through a mental imagery activity. They write down an exercise goal & are asked to practice the mental imagery twice a day for 3 weeks.
  * Participants take Baseline Survey 2.
  * Participants receive text messages reminding them to practice the mental imagery twice daily for 5 minutes each time (3 texts a week for 3 weeks).
  * Participants take surveys via text at the end of each week for 4 weeks.
  * 90 days post-baseline, participants complete a survey sent through the mail.
  * Participants may be contacted for another survey 1 year later.
  Interventions: Behavioral: Risk Assessment App; Other: Surveys; Behavioral: Audio Recording - Exercise; Other: Text message reminders; Other: Text Message Survey
- Risk Display Format:Text:Imagery Behavior:Sleep (Experimental): * With help from a research assistant, participants complete the Risk Assessment App. The App asks demographic & health questions. It then provides personalized risk estimates for participants' current activity level & how it would change with regular exercise.
  * Participants take Baseline Survey 1.
  * Participants listen to an audio recording that guides them through a mental imagery activity. They write down a sleep goal & are asked to practice the mental imagery twice a day for 3 weeks.
  * Participants take Baseline Survey 2.
  * Participants receive text messages reminding them to practice the mental imagery twice daily for 5 minutes each time (3 texts a week for 3 weeks).
  * Participants take surveys via text at the end of each week for 4 weeks.
  * 90 days post-baseline, participants complete a survey sent through the mail.
  * Participants may be contacted for another survey 1 year later.
  Interventions: Behavioral: Risk Assessment App; Behavioral: Audio Recording - Sleep; Other: Surveys; Other: Text message reminders; Other: Text Message Survey

INTERVENTIONS:
Behavioral: Risk Assessment App — The App provides participants with personalized risk results for colon cancer, breast cancer (women), heart disease, diabetes, and stroke.
Behavioral: Audio Recording - Sleep — -Participants imagine themselves improving sleep hygiene
  Arms: Risk Display Format:Risk Ladder:Imagery Behavior:Sleep; Risk Display Format:Table: Imagery Behavior:Sleep; Risk Display Format:Text:Imagery Behavior:Sleep
Other: Surveys — Assesses information comprehension, intentions, perceived risk and severity worry, self- efficacy, response efficacy, affect, race, education, age, numeracy, graph literacy, and exercise and sleep behaviors.
Behavioral: Audio Recording - Exercise — Participants imagine themselves improving exercise
  Arms: Risk Display Format:Risk Ladder:Imagery Behavior:Exercise; Risk Display Format:Table:Imagery Behavior:Exercise; Risk Display Format:Text:Imagery Behavior:Exercise
Other: Text message reminders — -Reminders to practice mental imagery
Other: Text Message Survey — -Assesses exercise behavior, intentions, actions plans, self-efficacy, affect, imagery vividness, and practice.

SUMMARY:
Epidemiology seeks to improve public health by identifying risk factors for cancer and other diseases and conveying that information to relevant audiences (e.g., physicians, the public). The audience is presumed to understand and use that information to make appropriate decisions about lifestyle behaviors and medical treatments. Yet, even though a single risk factor can affect the risk of multiple health outcomes, this information is seldom communicated to people in a way that optimizes their understanding of the importance of engaging in a single healthy behavior. Providing individuals with the ability to understand how a single behavior (obtaining sufficient physical activity) could affect their risk of developing multiple diseases could foster a more coherent and meaningful picture of the behavior's importance in reducing health risks, increase motivation and intentions to engage in the behavior, and over time improve public health.

The proposed study translates epidemiological data about five diseases that cause significant morbidity and mortality (i.e., colon cancer, breast cancer (women), heart disease, diabetes, and stroke) into a visual display that conveys individualized risk estimates in a comprehensible, meaningful, and useful way to diverse lay audiences.

ELIGIBILITY:
Inclusion Criteria:

* 30-64 years of age
* Less than (3) relevant comorbidities (diabetes, heart disease, stroke, and cancer, where cancer counts as (2) comorbidities for women but (1) for men)
* Having a SMS capable mobile phone that is not shared with anyone else

Exclusion Criteria:

* Not meeting national guidelines for aerobic physical activity (i.e., at least 150 minutes per week of moderate intensity aerobic physical activity)
* Participants from HRPO# 201501028 will be ineligible for this study
* Uses text messaging less than once per month

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 554 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Waters, MPH, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Risk Display Format:Risk Ladder:Imagery Behavior:Exercise | Risk Display Format:Risk Ladder:Imagery Behavior:Sleep | Risk Display Format:Table:Imagery Behavior:Exercise | Risk Display Format:Table: Imagery Behavior:Sleep | Risk Display Format:Text:Imagery Behavior:Exercise | Risk Display Format:Text:Imagery Behavior:Sleep
Started | 93 | 90 | 91 | 90 | 95 | 95
Completed | 80 | 78 | 85 | 84 | 88 | 85
Not Completed | 13 | 12 | 6 | 6 | 7 | 10
Not completed — Determined to be ineligible | 10 | 12 | 6 | 6 | 5 | 10
Not completed — Baseline data collection issues | 3 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Risk Display Format:Table:Imagery Behavior:Sleep; Risk Display Format:Text:Imagery Behavior:Sleep: * With help from a research assistant, participants complete the Risk Assessment App. The App asks demographic & health questions. It then provides personalized risk estimates for participants' current activity level & how it would change with regular exercise.
  * Participants take Baseline Survey 1.
  * Participants listen to an audio recording that guides them through a mental imagery activity. They write down a sleep goal & are asked to practice the mental imagery twice a day for 3 weeks.
  * Participants take Baseline Survey 2.
  * Participants receive text messages reminding them to practice the mental imagery twice daily for 5 minutes each time (3 texts a week for 3 weeks).
  * Participants take surveys via text at the end of each week for 4 weeks.
  * 90 days post-baseline, participants complete a survey sent through the mail.
  * Participants may be contacted for another survey 1 year later.
- Total: Total of all reporting groups
Arm/Group | Risk Display Format:Risk Ladder:Imagery Behavior:Exercise | Risk Display Format:Risk Ladder:Imagery Behavior:Sleep | Risk Display Format:Table:Imagery Behavior:Exercise | Risk Display Format:Table:Imagery Behavior:Sleep | Risk Display Format:Text:Imagery Behavior:Exercise | Risk Display Format:Text:Imagery Behavior:Sleep | Total
Number analyzed (Participants) | 80 | 78 | 85 | 84 | 88 | 85 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (9.8) | 47.3 (8.7) | 50.3 (9.9) | 49.8 (9.9) | 46.8 (10.7) | 47.2 (10.5) | 48.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 67 | 68 | 67 | 69 | 73 | 407
  Male | 17 | 11 | 17 | 17 | 19 | 12 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 1 | 5 | 4 | 2 | 17
  Not Hispanic or Latino | 76 | 77 | 84 | 79 | 84 | 83 | 483
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 1 | 0 | 1 | 0 | 0 | 0 | 2
  Asian/Pacific Islander | 1 | 0 | 2 | 0 | 1 | 2 | 6
  Black/African American | 27 | 35 | 26 | 37 | 37 | 23 | 185
  White/Caucasian | 49 | 43 | 50 | 40 | 46 | 56 | 284
  Multiracial/Other | 2 | 0 | 6 | 7 | 4 | 4 | 23
Region of Enrollment [Number; unit: participants]
  United States | 80 | 78 | 85 | 84 | 88 | 85 | 500
Vocational-technical training or less [Count of Participants; unit: Participants] | 20 | 20 | 14 | 14 | 15 | 14 | 97
Body mass index (BMI) - Obese [Count of Participants; unit: Participants] — -Having a BMI of 30 or greater
  Participants | 38 | 32 | 46 | 52 | 48 | 42 | 258
Body mass index (BMI) - Overweight [Count of Participants; unit: Participants] — -Having a BMI of 25 - less than 30
  Participants | 21 | 23 | 19 | 15 | 24 | 25 | 127
1+ comorbidity [Count of Participants; unit: Participants] — -Does the participant have one more serious comorbidities (cancer, diabetes, heart disease, stroke)?
  Participants | 14 | 6 | 21 | 17 | 19 | 15 | 92
Baseline Exercise (minutes per week in last 7 days) [Mean (Standard Deviation); unit: minutes] | 56.7 (44.8) | 56.9 (45.1) | 53.9 (47.4) | 50.2 (45.4) | 41.3 (41.1) | 56.0 (43.4) | 52.3 (44.7)
Self-Reported Health [Mean (Standard Deviation); unit: units on a scale] — -Self-reported health consisted of question asking "In general, would you say that your health is." with choices of Excellent, Very good, Good, Fair, or Poor. Measured on a scale of 1-5, with 5 being higher self-reported health.
  units on a scale | 3.0 (1.0) | 3.1 (0.9) | 3.0 (1.0) | 3.1 (0.9) | 3.0 (0.9) | 3.0 (0.9) | 3.0 (0.9)
Numeracy [Mean (Standard Deviation); unit: units on a scale] — * Scale of 0-3; Measured as a sum score of (correct/incorrect) of 3 questions, participant answers each question as fill in the blank.
  * "Imagine that we flip a fair coin 1,000 times. What is your best guess about how many times the coin would come up heads in 1,000 flips?"
  * "Image that the chance of getting a disease is 1%. If there were 1,000 people, about how many would be expected to get the disease?"
  * "Image that the chance of getting an infection is 1 in 1,000. What percent of people would be expected to get the infection?"
  units on a scale | 1.6 (1.0) | 1.3 (0.9) | 1.7 (1.0) | 1.5 (1.1) | 1.5 (1.1) | 1.6 (1.0) | 1.5 (1.0)
Graph literacy [Mean (Standard Deviation); unit: units on a scale] — * Scale of 1-4; Measured as a sum score of (correct/incorrect) of 4 questions. An example item is:
  * "The graph below shows the percentage of people who die from different types of cancer. About what percentage of people who die from cancer die from cancer B, cancer C, and cancer D combined?"
  units on a scale | 2.5 (1.1) | 2.1 (1.2) | 2.2 (1.2) | 2.3 (1.1) | 2.2 (1.2) | 2.6 (1.0) | 2.3 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 90-day Follow-up in Self Reported Weekly Minutes of Exercise
Time Frame: Baseline and up to 90 days
Population: Additional participants who did not complete the 90 day follow up survey or completed the survey over 8 weeks late, were inattentive responders, had text messaging errors, or were considered an outlier (>99th percentile) in change in minutes of exercise per week were excluded for analysis
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Risk Display Format:Risk Ladder:Imagery Behavior:Exercise | Risk Display Format:Risk Ladder:Imagery Behavior:Sleep | Risk Display Format:Table:Imagery Behavior:Exercise | Risk Display Format:Table: Imagery Behavior:Sleep | Risk Display Format:Text:Imagery Behavior:Exercise | Risk Display Format:Text:Imagery Behavior:Sleep
Number analyzed (Participants) | 70 | 66 | 72 | 67 | 73 | 72
minutes | 92.2 (12.7) | 37.5 (13.4) | 63.1 (12.4) | 60.0 (12.9) | 50.1 (12.5) | 49.3 (13.0)
Statistical Analysis 1: Comparison: Risk Display Format:Risk Ladder:Imagery Behavior:Sleep vs Risk Display Format:Table: Imagery Behavior:Sleep vs Risk Display Format:Text:Imagery Behavior:Sleep; The investigators tested whether weekly minutes of exercise at 90 day follow-up was higher in the exercise mental imagery condition than in the sleep mental imagery condition; Test type: Superiority — A Dunnett adjustment was used to adjust for multiple comparisons; p = 0.0288, ANCOVA; Covariates: sex, race, age, education, health literacy, season, risk display problem, acceptability, self-reported health, and baseline exercise
Statistical Analysis 2: Comparison: Risk Display Format:Text:Imagery Behavior:Exercise vs Risk Display Format:Text:Imagery Behavior:Sleep; -The investigators tested whether weekly minutes of exercise differed among the three risk display formats: risk ladder, table, and alphanumeric text; Test type: Superiority — -A Dunnett adjustment was used to adjust for multiple comparisons; p = 0.3329, ANCOVA; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Risk Display Format:Text:Imagery Behavior:Sleep; -The investigators tested whether weekly minutes of exercise was influenced by an interaction between risk display format and mental imagery behavior; Test type: Superiority — -A Dunnett adjustment was used to adjust for multiple comparisons; p = 0.0215, ANCOVA; [statistical method as in outcome 1, analysis 1]

2. Primary Outcome: Difference in Gist Comprehension of Risk Information by Risk Display Format
Description: * Risk display format = risk ladder, table, or text
  * Gist comprehension of risk information: being able to extract the bottom-line meaning of information provided by the website (e.g., if exercising decreased heath risk)
  * Measured by the sum of (4) questions coded as correctly comprehending risk information (1 point) or incorrectly comprehending risk information (0 points), with a total score range of 0=low comprehension to 4=high comprehension. Higher comprehension is considered a better outcome.
  * All comprehension questions have an additional "don't know" option, which is counted as incorrect.
  * To limit participant burden, the investigators assessed comprehension for diabetes only, instead of all diseases as planned.
  * Comprehension will not be assessed for people who report a history of diabetes because they are not given risk information.
Time Frame: Baseline
Population: This study was designed as a 3X2 factorial design & only the risk display format intervention (risk ladder, table, or text) was looked at for this outcome, as participants had not yet received the mental imagery intervention, thus it could not affect this outcome.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Risk Display Format: Risk Ladder: -The personalized risk estimates were shown to participants as a risk ladder.
- Risk Display Format: Table: -The personalized risk estimates were shown to participants as a table.
- Risk Display Format: Text: -The personalized risk estimates were shown to participants as text.
Arm/Group | Risk Display Format: Risk Ladder | Risk Display Format: Table | Risk Display Format: Text
Number analyzed (Participants) | 125 | 120 | 127
score on a scale | 3.6 (0.1) | 3.4 (0.1) | 3.2 (0.1)
Statistical Analysis 1: Comparison: Risk Display Format: Risk Ladder vs Risk Display Format: Table vs Risk Display Format: Text; -This study was designed as a 3X2 factorial design and only the risk display format intervention (risk ladder, table, or text) was looked at for this outcome, as participants had not yet received the mental imagery intervention, thus it could not affect this outcome. A Dunnett adjustment was used to adjust for multiple comparisons; Test type: Superiority; p = 0.0333, ANCOVA — -A Dunnett adjustment was used to adjust for multiple comparisons; Covariates were sex, race, age, education, numeracy, and graph literacy

3. Primary Outcome: Difference in Verbatim Comprehension of Risk Information by Risk Communication Strategy
Description: * Risk communication strategy = risk ladder, table, or text
  * Verbatim comprehension of risk information: being able to recall the exact information specific to diabetes risk and hours of recommended weekly physical activity
  * Measured by the sum of (3) questions coded as correctly comprehending information (1 point) or incorrectly comprehending information (0 points), with a total score range of 0=low comprehension to 3=high comprehension. Higher comprehension is considered a better outcome.
  * All comprehension questions have an additional "don't know" option, which is counted as incorrect.
  * To limit participant burden, the investigators assessed comprehension for diabetes only, instead of all diseases as planned.
  * Comprehension will not be assessed for people who report a history of diabetes because they are not given risk information.
Time Frame: Baseline
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risk Display Format: Risk Ladder | Risk Display Format: Table | Risk Display Format: Text
Number analyzed (Participants) | 125 | 120 | 127
score on a scale | 1.6 (0.1) | 1.6 (0.1) | 1.5 (0.1)
Statistical Analysis 1: Comparison: Risk Display Format: Risk Ladder vs Risk Display Format: Table vs Risk Display Format: Text; This study was designed as a 3X2 factorial design & only the risk display format intervention (risk ladder, table, or text) was looked at for this outcome, as participants had not yet received the mental imagery intervention, thus it could not affect this outcome; Test type: Superiority; p = 0.4946, ANCOVA — -A Dunnett adjustment was used to adjust for multiple comparisons; Covariates were sex, race, age, education, numeracy, and graph literacy

4. Primary Outcome: Difference in Self-reported Intentions to Engage in Physical Activity by Risk Display Format
Description: * Risk display format = risk ladder, table, or text
  * Self-reported physical activity intentions is defined as intentions to engage in physical activity in the next 3 months
  * Measured as an average of three variables, each measured on a 5 point Likert Scale (range: 1=lower intentions to 5=higher intentions)
  * Higher intentions are considered a better outcome
Time Frame: Baseline
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Risk Display Format: Risk Ladder | Risk Display Format: Table | Risk Display Format: Text
Number analyzed (Participants) | 125 | 120 | 127
score on a scale | 3.9 (0.1) | 4.0 (0.1) | 3.8 (0.1)
Statistical Analysis 1: Comparison: Risk Display Format: Risk Ladder vs Risk Display Format: Table vs Risk Display Format: Text; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1397, ANCOVA; Covariates were sex, race, age, education, numeracy, and graph literacy

5. Secondary Outcome: Effect of the Intervention on Physical Activity Levels as Measured by Maintenance Self-efficacy
Description: * Maintenance Self-efficacy is defined as being sure one can engage in physical activity even when it is hard
  * Measured on a 4 point Likert Scale (range: 1=lower Maintenance Self-efficacy to 4=higher Maintenance Self-efficacy)
  * Higher maintenance self-efficacy is considered a better outcome
  * Note: to limit participant burden, the investigators used a single item instead of averaging across multiple items
Time Frame: 90 days
Population: Due to the limitations of data collection & concerns about overburdening participants with too many survey questions, the investigators only assessed exercise-related maintenance self-efficacy among participants who engaged in the exercise-related mental imagery condition.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Mental Imagery Behavior: Exercise: -Participants engaged in mental imagery related to exercise goals
Arm/Group | Mental Imagery Behavior: Exercise
Number analyzed (Participants) | 229
score on a scale | 2.95 (0.05)
Statistical Analysis 1: Comparison: Mental Imagery Behavior: Exercise; The secondary outcomes are hypothesized mediators of the effect of exercise-related mental imagery activities on future exercise behavior (e.g., exercise mental imagery will increase future exercise behavior by increasing exercise maintenance self-efficacy). Because these analyses are relevant only for the exercise condition, and the dichotomous mental imagery variable includes both exercise and sleep, it is not appropriate to include the dichtomous mental imagery variable in this analysis; Test type: Superiority; p = 0.0070, Mixed Models Analysis — Covariates: sex, race, age, education, risk display issue, health literacy, season, acceptability, self-reported health, adherence, baseline exercise

6. Secondary Outcome: Effect of the Intervention on Physical Activity Levels as Measured by Recovery Self-efficacy
Description: * Recovery Self-efficacy is defined as being sure one can re-engage in physical activity after putting it off
  * Measured on a 4 point Likert Scale (range: 1=lower recovery Self-efficacy to 4=higher recovery Self-efficacy)
  * Higher recovery self-efficacy is considered a better outcome
  * Note: to limit participant burden, the investigators used a single item instead of averaging across multiple items
Time Frame: 90 days
Population: Due to the limitations of data collection & concerns about overburdening participants with too many survey questions, the investigators only assessed exercise-related recovery self-efficacy among participants who engaged in the exercise-related mental imagery condition.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mental Imagery Behavior: Exercise
Number analyzed (Participants) | 229
score on a scale | 3.26 (0.05)
Statistical Analysis 1: Comparison: Mental Imagery Behavior: Exercise; The secondary outcomes are hypothesized mediators of the effect of exercise-related mental imagery activities on future exercise behavior (e.g., exercise mental imagery will increase future exercise behavior by increasing exercise recovery self-efficacy). Because these analyses are relevant only for the exercise condition, and the dichotomous mental imagery variable includes both exercise and sleep, it is not appropriate to include the dichtomous mental imagery variable in this analysis; Test type: Superiority; p = 0.8793, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

7. Secondary Outcome: Effect of the Intervention on Physical Activity Levels as Measured by Affective Attitudes to Exercise - Enjoying Behavior
Description: * Affective Attitudes to Exercise - Enjoying Behavior is defined as thinking getting regular exercise is enjoyable
  * Measured on a 4 point Likert Scale (range: 1=lower Affective Attitudes to Exercise to 4=higher Affective Attitudes to Exercise)
  * Higher Affective Attitudes to Exercise - Enjoying Behavior is considered a better outcome
  * Note: to limit participant burden, the investigators used a single item instead of averaging across multiple items
Time Frame: 90 days
Population: Due to the limitations of data collection and concerns about overburdening participants with too many survey questions, the investigators only assessed exercise-related affective attitudes among participants who engaged in the exercise-related mental imagery condition.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mental Imagery Behavior: Exercise
Number analyzed (Participants) | 229
score on a scale | 3.05 (0.05)
Statistical Analysis 1: Comparison: Mental Imagery Behavior: Exercise; The secondary outcomes are hypothesized mediators of the effect of the exercise-related mental imagery activities on future exercise behavior (e.g., exercise mental imagery will increase future exercise behavior by increasing exercise affective attitudes). Because these analyses are relevant only for the exercise condition, and the dichotomous mental imagery variable includes both exercise and sleep, it is not appropriate to include the dichotomous mental imagery variable in this analysis; Test type: Superiority; p = 0.4673, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

8. Secondary Outcome: Effect of the Intervention on Physical Activity Levels as Measured by Affective Attitudes to Exercise - Thinking Behavior is Unpleasant
Description: * Affective Attitudes to Exercise - Thinking Behavior is Unpleasant is defined as not thinking getting regular exercise is unpleasant
  * Measured on a 4 point Likert Scale (range: 1=lower Affective Attitudes to Exercise to 4=higher Affective Attitudes to Exercise)
  * Higher Affective Attitudes to Exercise - Thinking Behavior is Unpleasant is considered a better outcome
  * Note: to limit participant burden, the investigators used a single item instead of averaging across multiple items
Time Frame: 90 days
Population: as for outcome 7
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mental Imagery Behavior: Exercise
Number analyzed (Participants) | 229
score on a scale | 3.19 (0.05)
Statistical Analysis 1: Comparison: Mental Imagery Behavior: Exercise; The secondary outcomes are hypothesized mediators of the effect of the exercise-related mental imagery activities on future exercise behavior (e.g., exercise mental imagery will increase future exercise behavior by increasing exercise unpleasant feelings). Because these analyses are relevant only for the exercise condition, and the dichotomous mental imagery variable includes both exercise and sleep, it is not appropriate to include the dichotomous mental imagery variable in this analysis; Test type: Superiority; p = 0.1916, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

9. Secondary Outcome: Effect of the Intervention on Physical Activity Levels as Measured by Perceived Vividness of Self-regulatory Imagery
Description: * Perceived Vividness of Self-regulatory Imagery is defined as having clear and vivid images of steps towards getting physical activity
  * Measured as an average of two variables measured on a 4 point Likert Scale (range: 1=lower Perceived Vividness of Self-regulatory Imagery to 4=higher Perceived Vividness of Self-regulatory Imagery)
  * Higher Perceived Vividness of Self-regulatory Imagery is considered a better outcome
  * Note: to limit participant burden, the investigators used a single item instead of averaging across multiple items
Time Frame: 90 days
Population: Due to the limitations of data collection and concerns about overburdening participants with too many survey questions, the investigators only assessed exercise-related perceived vividness of self-regulatory imagery among participants who engaged in the exercise-related mental imagery condition.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mental Imagery Behavior: Exercise
Number analyzed (Participants) | 229
score on a scale | 3.36 (0.04)
Statistical Analysis 1: Comparison: Mental Imagery Behavior: Exercise; The secondary outcomes are hypothesized mediators of the effect of the exercise-related mental imagery activities on future exercise behavior (e.g., exercise mental imagery will increase future exercise behavior by increasing exercise imagery vividness). Because these analyses are relevant only for the exercise condition, and the dichotomous mental imagery variable includes both exercise and sleep, it is not appropriate to include the dichotomous mental imagery variable in this analysis; Test type: Superiority; p = 0.8661, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

10. Secondary Outcome: Effect of the Intervention on Physical Activity Levels as Measured by Action Planning
Description: * Action planning is defined as having a detailed plan about getting adequate physical activity
  * Measured as an average of three variables measured on a 4 point Likert Scale (range: 1=lower action planning to 4=higher action planning)
  * Higher action planning is considered a better outcome
  * Note: to limit participant burden, the investigators used a single item instead of averaging across multiple items
Time Frame: 90 days
Population: Due to the limitations of data collection and concerns about overburdening participants with too many survey questions, the investigators only assessed exercise-related action planning among participants who engaged in the exercise-related mental imagery condition.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mental Imagery Behavior: Exercise
Number analyzed (Participants) | 229
score on a scale | 3.52 (0.03)
Statistical Analysis 1: Comparison: Mental Imagery Behavior: Exercise; The secondary outcomes are hypothesized mediators of the effect of the exercise-related mental imagery activities on future exercise behavior (e.g., exercise mental imagery will increase future exercise behavior by increasing exercise action planning). Because these analyses are relevant only for the exercise condition, and the dichotomous mental imagery variable includes both exercise and sleep, it is not appropriate to include the dichotomous mental imagery variable in this analysis; Test type: Superiority; p = 0.0711, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

11. Secondary Outcome: Effect of the Intervention on Physical Activity Levels as Measured by Coping Planning
Description: * Coping planning is defined as having a detailed plan of solving problems that may prevent getting adequate physical activity
  * Measured on a 4 point Likert Scale (range: 1=lower Coping Planning to 4=higher Coping Planning)
  * Higher coping planning is considered a better outcome
  * Note: to limit participant burden, the investigators used a single item instead of averaging across multiple items
Time Frame: 90 days
Population: Due to the limitations of data collection and concerns about overburdening participants with too many survey questions, the investigators only assessed exercise-related coping planning among participants who engaged in the exercise-related mental imagery condition.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mental Imagery Behavior: Exercise
Number analyzed (Participants) | 229
score on a scale | 2.98 (0.04)
Statistical Analysis 1: Comparison: Mental Imagery Behavior: Exercise; The secondary outcomes are hypothesized mediators of the effect of the exercise-related mental imagery activities on future exercise behavior (e.g., exercise mental imagery will increase future exercise behavior by increasing exercise coping planning). Because these analyses are relevant only for the exercise condition, and the dichotomous mental imagery variable includes both exercise and sleep, it is not appropriate to include the dichotomous mental imagery variable in this analysis; Test type: Superiority; p = 0.0365, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

12. Secondary Outcome: Effect of the Intervention on Physical Activity Levels as Measured by Action Self-efficacy
Description: * Action self-efficacy is defined as having the confidence to engage in physical activity
  * Measured on a 4 point Likert Scale (range: 1=lower Action Self-efficacy to 4=higher Action Self-efficacy)
  * Higher Action Self-efficacy is considered a better outcome
  * Note: to limit participant burden, the investigators used a single item instead of averaging across multiple items
Time Frame: 90 days
Population: Due to the limitations of data collection and concerns about overburdening participants with too many survey questions, the investigators only assessed exercise-related action self-efficacy among participants who engaged in the exercise-related mental imagery condition.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mental Imagery Behavior: Exercise
Number analyzed (Participants) | 229
score on a scale | 3.36 (0.04)
Statistical Analysis 1: Comparison: Mental Imagery Behavior: Exercise; The secondary outcomes are hypothesized mediators of the effect of the exercise-related mental imagery activities on future exercise behavior (e.g., exercise mental imagery will increase future exercise behavior by increasing exercise action self-efficacy). Because these analyses are relevant only for the exercise condition, and the dichotomous mental imagery variable includes both exercise and sleep, it is not appropriate to include the dichotomous mental imagery variable in this analysis; Test type: Superiority; p = 0.1511, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for this study.
Description: Adverse events were not collected for this study.
Arm/Group | Risk Display Format:Risk Ladder:Imagery Behavior:Exercise | Risk Display Format:Risk Ladder:Imagery Behavior:Sleep | Risk Display Format:Table:Imagery Behavior:Exercise | Risk Display Format:Table:Imagery Behavior:Sleep | Risk Display Format:Text:Imagery Behavior:Exercise | Risk Display Format:Text:Imagery Behavior:Sleep
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/78 | 0/85 | 0/84 | 0/88 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT03255291/Prot_SAP_000.pdf